CLINICAL TRIAL: NCT01892670
Title: Storage Temperature and Quality of Leucoreduced Whole Blood
Acronym: BFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian Armed Forces Medical Service (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/2279
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2017-08

CONDITIONS: Trauma; Austere Environment; Blood Bank; Buddy Transfusion
Keywords: Blood; Whole blood; Cold-storage; Filtration; Transfusion; Platelet-function
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Filtered whole blood (Experimental): Leukocyte-reduced whole blood, 2 hours holding-time after collection. Gravitational filtration.
  Device: Terumo IMUFLEX WB(Whole blood)-SP(saving platelets) collection bag system
  Interventions: Other: Donation of 1 whole blood unit
- Unfiltered whole blood (Experimental): Non-leukocyte-reduced whole blood, 2 hours holding-time after collection.
  Device: Terumo IMUFLEX WB-SP collection bag system
  Interventions: Other: Donation of 1 whole blood unit
- Warm-filtered whole blood (Experimental): Leukocyte-reduced whole blood, no holding-time after collection. Gravitational filtration.
  Device: Terumo IMUFLEX WB-SP collection bag system
  Interventions: Other: Donation of 1 whole blood unit
- Forced warm-filtration of whole bood (Experimental): Leukocyte-reduced whole blood, no holding-time after collection. Forced filtration.
  Device: Terumo IMUFLEX WB-SP collection bag system
  Interventions: Other: Donation of 1 whole blood unit
- RCC produced from cold-stored whole blood (Experimental): RCC production from 7 days old, cold-stored, leukocyte-reduced whole blood. Units stored for another 35 days. (42 days of storage in total).
  Devices: Terumo IMUFLEX WB-SP/WB-RP collection bag systems.
  Interventions: Other: Donation of 1 whole blood unit
- RCC produced from cold-stored non-filtered whole blood (Experimental): RCC production from 7 days old, cold-stored, non-leukocyte-reduced whole blood. Units stored for another 35 days. (42 days of storage in total).
  Devices: Terumo IMUFLEX WB-SP/WB-RP(removing platelets) collection bag systems.
  Interventions: Other: Donation of 1 whole blood unit

INTERVENTIONS:
Other: Donation of 1 whole blood unit — Donation of 450-500 mL of whole blood according to local blood bank procedures and national guidelines.
  Other Names: Terumo IMUFLEX WB-SP collection bag system.

SUMMARY:
In a combat situation the need for safe and high-quality blood products is increasing. WB (Whole Blood) is used in many trauma situations, but we wish to investigate whether there is an even better whole blood product.

The purpose of this study is to examine the quality of leucoreduced, cold-stored whole blood. We also wish to examine the effects of filtration of whole blood without a 1-2 hour holding-time (warm-filtration) and the effects of forced filtration. We also wish to explore the possibility of using cold-stored WB for production of RCC.

Analyses are performed with a main focus to investigate function and quality of red blood cells and platelets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age between 18 and 70
* Negative pregnancy test (women in fertile age)
* Blood pressure range: (160-100)/(100-40)
* Pulse range: 40-100

Exclusion Criteria:

* Usage of platelet-influencing medication
* Mild flu or more severe illnesses
* Open wound
* Pregnancy or trying to get pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Platelet function | After 10 days of cold-storage
  Platelet function is assessed by various parameters, such as thrombelastography (TEG), Multiplate and flow cytometry (Lactadherin, Calcein violet AM, ++).

SECONDARY OUTCOMES:
Leukocyte count | After leukocyte filtration
  Filtered whole blood should have a concentration less than 1*10^6 cells/L to avoid transfusion reactions.

OTHER OUTCOMES:
Hemolysis | After 42 days of storage
  RCC should not have a hemolysis of more than 0.8 %. We investigate this up to 42 days (35 days as RCC) (arm 5 +6)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Strandenes, MD, Principal Investigator — Haukeland University Hospital and Norwegian Naval Special Operation Commando
Locations (1):
- Haukeland University Hospital, Dept of Immunology and Transfusion Medicine, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No